CLINICAL TRIAL: NCT00751244
Title: Breaking the Cycle for Women With Behavioral Problems and Crime
Brief Title: Mothers Overcoming and Managing Stress
Acronym: MOMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: U.S. Department of Justice (U.S. Federal Agency)
Responsible Party: Julian Ford, Ph.D., University of Connecticut Health Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-051H-1; 2004-DD-BX-1025
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2010-09-27 (Estimated); Status verified 2010-09

CONDITIONS: Posttraumatic Stress Disorder; PTSD
Keywords: women; posttraumatic stress disorder; PTSD; psychotherapy; clinical trial; emotion regulation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Emotional Regulation | interventions — Educational Status; Therapeutics; Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): 12 weekly sessions of one-to-one TARGET (psychotherapy)
  Interventions: Behavioral: Trauma Affect Regulation: Guide for Education and Therapy
- 2 (Active Comparator): 12 weekly sessions of one-to-one PCT (psychotherapy)
  Interventions: Behavioral: Present Centered Therapy (PCT) - psychotherapy
- 3 (Other): 90-day wait-list group
  Interventions: Other: No-treatment "waitlist" group

INTERVENTIONS:
Behavioral: Trauma Affect Regulation: Guide for Education and Therapy — Trauma Affect Regulation: Guide for Education and Therapy (TARGET; Ford & Russo, 2006) is a manualized gender-specific treatment for PTSD. TARGET teaches a practical 7-step sequence of skills for processing and managing trauma-related reactions to current stressful experiences, summarized by a mnemonic ("FREEDOM"), e.g., Focusing ("F"), Recognizing current triggers. TARGET also involves creative arts activities, i.e., personalized "lifelines" via collage, drawing, poetry, and writing that may include traumatic experiences but emphasize "life story" narrative reconstruction with no exposure therapy.
  Other Names: Julian Ford
  Arms: 1
Behavioral: Present Centered Therapy (PCT) - psychotherapy — Present Centered Therapy (PCT) is a 12-session supportive therapy adapted a 14-session version co-developed by the first author (McDonagh-Coyle et al., 2005). Psychoeducation is provided about the link between traumatic events, PTSD symptoms, and problems in relationships, and social problem solving skills are taught to address the "traumagenic dynamics" of betrayal, stigma, powerlessness, and sexualization (Finkelhor, 1987). PCT focuses on addressing current problems rather than trauma memory-based exposure therapy, and uses a distinctive mnemonic to organize the skill set. PCT has clients keep a journal of relational stressors and responses as between-session homework.
  Other Names: McDonagh-Coyle
  Arms: 2
Other: No-treatment "waitlist" group — After a 90 day wait-list period, participants were invited to choose one of the treatment approaches (PCT or TARGET) and engage in 12 sessions of therapy.
  Arms: 3

SUMMARY:
The study is a randomized trial of two manualized 12-session one-to-one educational and therapeutic interventions for post-traumatic stress disorder (PTSD), to test and compare their efficacy for reducing PTSD symptoms as a means of prevention of intergenerational victimization by or involvement in criminal activities with at-risk mothers. The two therapies are (1) Trauma Affect Regulation: Guide for Education and Therapy (TARGET) and (2) Present Centered Therapy (PCT). The study also included a wait-list comparison condition in which participants were offered one of the two therapies following completion of baseline and posttest assessments.

DETAILED DESCRIPTION:
Hypotheses, Objectives and Aims:

The study is a randomized clinical trial comparing two stress management counseling interventions with a wait-list comparison condition to determine their efficacy in addressing behavioral, cognitive, affective, and interpersonal effects of PTSD that often occurs for persons living in adverse socioeconomic circumstances and in violent families and communities. One goal of the study is to reduce the severity of or produce remission from PTSD, in order to reduce impulsivity, aggression, dissociation, and isolation by high-risk or previously incarcerated women. The long-term goal, which will be assessed in subsequent studies over time is to reduce the likelihood of their or their children becoming involved in, or victimized by other persons' involvement in, illegal activities. Children will not be involved in the present study, only women who are the mothers of young children.

Aim #1: To test the efficacy of TARGET and PCT. TARGET (Frisman, L., Ford, J. D., Lin, H., Mallon, S., & Chang, R., 2008) and PCT (McDonagh A, Friedman M, McHugo G, Ford J, Sengupta A, Mueser K, Demment CC, Fournier D, Schnurr PP, Descamps M., 2005) have demonstrated efficacy in randomized trial studies, but have not been tested specifically with mothers of young children. The study will assess outcomes that are of potential importance not only for the well being of the participating women but for their ability to develop secure attachments with their child which are protective against exposure to violence, crime, and victimization and associated with positive psychosocial development by children. Outcome measures reflect self-regulatory capacities compromised by trauma that are essential for effective caregiving by adults.

Aim #2: To compare the efficacy of TARGET and PCT on theory-based differential outcomes. TARGET and PCT use similar but different therapeutic strategies. Each teaches skills for managing negative emotions and critical symptoms (e.g., inhibiting impulsivity). TARGET teaches a skill sequence for affect regulation and social/interoceptive information processing, while PCT teaches a skill sequence for recognizing and solving problems in relationships. We expect that TARGET and PCT will reduce stress-related avoidance and depression and enhance active coping with current stressors. TARGET should be superior to PCT in enhancing the ability to cope with trauma memories, stress reactivity, and anxiety, and therefore the ability to remain free from illegal activities or future or further involvement with criminal justice systems. PCT should be superior to TARGET in enhancing the participant's overall social adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-50 years old (or emancipated minor)
* Primary care-giver of a child aged 0-5 years old
* A history of incarceration, or substance abuse, or exposure to violence
* Mentally able to participate and provide valid consent
* Able to complete the consent process, interviews, self-report measure and treatment/intervention primarily in English
* Willing to consent to be audio and/or videotaped for research purposes in intervention sessions
* Current post-traumatic stress disorder as assessed by study personnel

Exclusion Criteria:

* Imminently suicidal
* Past 30 days inpatient psychiatric treatment

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2005-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Reduced PTSD symptoms/impairment as evidenced by improvements on the Clinician Administered PTSD Scale (CAPS), Post-Traumatic Cognitions Inventory (PTCI), Traumatic Memories Questionnaire (TMQ), and the Interpretation of PTSD Symptoms Inventory (IPSI). | post-therapy, 3-month and 6-month follow-ups

SECONDARY OUTCOMES:
Improved affect/interpersonal self-regulation as evidenced by improvement on the Negative Mood Regulation Scale, Inventory of Interpersonal Problems, Multiscale Dissociation Inventory, Anxiety Inventory, and Beck Depression Inventory. | Post-treatment, 3-month and 6-month follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Julian Ford, Ph.D., Principal Investigator — UConn Health; Joan Levine, M.P.H., Study Director — UConn Health
Locations (2):
- United States (2):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Burgdorf Clinic/Bank of America Health Center on the Mount Sinai Campus of Saint Francis Hospital and Medical Center, Hartford, Connecticut

REFERENCES:
- [Background] Finkelhor, D. (1987). The trauma of child sexual abuse. Journal of Interpersonal Violence, 2, 348-366.
- [Background] Ford JD, Russo E. Trauma-focused, present-centered, emotional self-regulation approach to integrated treatment for posttraumatic stress and addiction: trauma adaptive recovery group education and therapy (TARGET). Am J Psychother. 2006;60(4):335-55. doi: 10.1176/appi.psychotherapy.2006.60.4.335. PMID 17340945
- [Background] McDonagh A, Friedman M, McHugo G, Ford J, Sengupta A, Mueser K, Demment CC, Fournier D, Schnurr PP, Descamps M. Randomized trial of cognitive-behavioral therapy for chronic posttraumatic stress disorder in adult female survivors of childhood sexual abuse. J Consult Clin Psychol. 2005 Jun;73(3):515-24. doi: 10.1037/0022-006X.73.3.515. PMID 15982149
- [Background] Ford, J. D. (2002). Traumatic victimization in childhood and persistent problems with oppositional-defiance. Journal of Trauma, Maltreatment, and Aggression, 11, 25-58.
- [Background] Wolpaw, J., Ford, J. D., Newman, E., Davis, J. L., & Briere, J. (2005). Trauma Symptom Checklist for Children: In T. Grisso, G. Vincent & D. Seagrave (Eds.), Mental health screening and assessment in juvenile justice (pp. 152-165). New York: Guilford.
- [Background] Frisman, L., Ford, J. D., Lin, H., Mallon, S., & Chang, R. (in press). Outcomes of trauma treatment using the TARGET model. Journal of Groups in Addiction and Recovery